CLINICAL TRIAL: NCT01653834
Title: Feasibility of Lymphocyte Reinfusion in Newly Diagnosed High Grade Gliomas
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J11162; NA_00068991 (Other: JHMIRB)
Record Dates: First submitted 2012-07-12; First posted 2012-07-31 (Estimated); Last update posted 2018-11-07 (Actual); Status verified 2018-11

CONDITIONS: Glioblastoma
Keywords: lymphopenia
MeSH Terms: conditions — Glioblastoma; Lymphopenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lymphocyte harvesting & reinfusion (Experimental): Patients with a newly diagnosed high grade glioma (Grade III or IV), have a post-operative treatment plan that includes standard radiation and temozolomide, and have normal bone marrow function with Hematocrit ≥ 30%, platelet ≥ 100K, ANC ≥ 1000, and absolute lymphocyte count ≥ 1000 prior entry to this study are eligible for enrollment.
  Interventions: Procedure: Lymphocyte harvesting & reinfusion

INTERVENTIONS:
Procedure: Lymphocyte harvesting & reinfusion — Lymphocytes will be collected and stored approximately one week prior to initiating concurrent radiation therapy (RT) and temozolomide (TMZ). Two lymphocyte collections are allowed. After the patient has completed 6 weeks of RT/TMZ, all of the collected lymphocytes will be re-infused. After lymphocyte re-infusion, Heme-8 and absolute lymphocyte count (ALC) will be checked per standard of care. The absolute increase in ALC as the primary endpoint will be assessed 4 weeks after lymphocyte re-infusion.

SUMMARY:
This research study is being done to see if lymphocytes can be collected from patients with high grade gliomas before they start standard radiation and chemotherapy. (Lymphocytes are cells that normally circulate in the blood and are an essential part of the immune system). The investigators goal is to store these and give them back to the patient after radiation is completed. This is part of a larger effort that will attempt to preserve the immune system from the effects of radiation and chemotherapy.

DETAILED DESCRIPTION:
The patients blood will be collected (apheresis) before starting the patients planned standard of care radiation therapy and chemotherapy:

* An IV will be inserted into the vein in the patients arm.
* The blood will be sent to a machine that removes the lymphocytes and returns the rest to the patient.
* This procedure will last from 1 hour and 15 minutes to 4 hours.
* During this time the patient will also be treated with a blood thinner to prevent the blood from clotting in the machine.
* The lymphocytes will be counted and stored. If an insufficient number were collected, we will ask for another similar collection in about 1 week.
* After the patient has completed the full 6 weeks of radiation, all of the lymphocytes will be returned to the patient through a simple intravenous infusion. A larger intravenous access (i.e. midline) might be needed. Any cells that are not reinfused will be stored for 1 year and then discarded.
* Study bloods (10 ml) will be collected at the time of lymphocyte collection, prior lymphocyte reinfusion, and then every 2 weeks until week 20th. These blood samples will be stored and used for future analysis.

Blood counts are obtained weekly as part of standard care for patients with this kind of brain tumor. For the first 14 weeks after the lymphocyte reinfusion we will be doing some extra tests on the routinely collected blood to see how the effective the reinfused lymphocytes are in raising the patients lymphocyte counts. These results will be available to the patients treating physician.

At no time will this study interfere with the patients planned standard of care radiation and chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* • Age≥18 year

  * New diagnosed high grade glioma
  * Post-operative treatment with standard RT/TMZ
  * Karnofsky performance status ≥ 60%
  * Normal bone marrow function with Hematocrit ≥ 30%, platelet ≥ 100K, ANC ≥ 1000, and absolute lymphocyte count ≥ 1000 prior entry to this study. Blood product transfusions are allowed.

Exclusion Criteria:

* Prior radiation therapy, chemotherapy, immunotherapy or therapy with biologic agents or hormonal therapy for their brain tumor are excluded. Glucocorticoid therapy is allowed.
* Fresh CNS bleed, current anticoagulation use; and anti-VEGF therapy in past 6 weeks are excluded.
* Patients must not have taken an ACE inhibitor within last 24 hours prior to apheresis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2012-07; Primary Completion 2014-01 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
the feasibility of lymphocyte harvesting and reinfusion | 10 weeks
  this will be considered a feasible approach if 5 of the 10 patients to be accrued have an absolute lymphocyte count increase of 300 cells per mm3 at 4 weeks after reinfusion.

SECONDARY OUTCOMES:
the number of lymphocytes that can be harvested in this pt population | 10 weeks
  the number of lymphocytes harvested per patient
duration of lymphocyte rise following lymphocyte reinfusion | 10 weeks
  how long will lymphocyte counts remain elevated after reinfusion
changes in lymphocyte subtypes following collection and reinfusion | 10 weeks
  changes in lymphocyte subtype between collection and reinfusion as a result of freezing for storage.

CONTACTS AND LOCATIONS:
Overall Officials: Stuart A Grossman, MD, Study Chair — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States